CLINICAL TRIAL: NCT00259558
Title: Prospektive, Randomisierte Doppelblinde Studie Zur Dosisfindung Von Intestinal Redardiert Freigesetztem Phosphatidylcholin Bei Chronisch Aktiver Pancolitis Ulcerosa
Brief Title: Dose Finding Study for Retarded Phosphatidylcholine in Pancolitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Prof. Wolfgang Stremmel (Unknown); Dietmar Hopp Stiftung (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC3; EC - L069/2003; BFARM - 402 2919
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2007-02-12 (Estimated); Status verified 2007-02

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Dose Finding; Phosphatidylcholine
MeSH Terms: conditions — Colitis, Ulcerative

INTERVENTIONS:
Drug: retarded release phosphatidylcholine

SUMMARY:
The purpose of this study is to find the optimal dose of retarded release Phosphatidylcholine in the most severe form of ulcerative colitis.

The hypothesis is that ulcerative colitis (UC) is caused by a barrier dysfunction of the colonic mucus layer. The background of the study is the finding, that the phosphatidylcholine (PC) content of the colonic mucus is strongly reduced in UC compared to healthy controls and patients with Crohn´s disease. The content was meuasured in non-inflamed areas of the colon in UC. Thus, we evaluate whether a substitution of colonic PC is an effective method.

DETAILED DESCRIPTION:
Design: prospective, randomized, double-blind, dose-finding study with retarded phosphatidylcholine.

Population: 10 patients per dose group (6 doses) - 60 patients Remark: this includes to historic groups from another study Inclusion criteria: Ulcerative Pancolitis with chronic active course and a clinical index (Rachmilewitz) over 7 and more, endoscopic index of at least 7 or more. No systemic steroids or immunosuppressants since 4 weeks.

Exclusion criteria: Pregnancy & fulminant course

ELIGIBILITY:
Inclusion Criteria:

* chronic active ulcerative pancolitis
* course more than 4 months
* clinical index rachmilewitz 7 or more
* endoskopic index 7 or more

Exclusion Criteria:

* steroids in the last 4 weeks
* immunosuppressants in the last 4 weeks
* use of topical klymsa
* pregnancy
* fulminant course
* infectious colitis

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-04; Study Completion 2006-03

PRIMARY OUTCOMES:
Absolute change in clinical activity index (Rachmilewitz).

SECONDARY OUTCOMES:
Secondary end points include >50% changes in clinical and endoscopic activity index (EAI).
Histology and life quality are reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Stremmel, Professor, Principal Investigator — University Heidelberg
Locations (1):
- Medical Hospital Unversity Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Stremmel W, Merle U, Zahn A, Autschbach F, Hinz U, Ehehalt R. Retarded release phosphatidylcholine benefits patients with chronic active ulcerative colitis. Gut. 2005 Jul;54(7):966-71. doi: 10.1136/gut.2004.052316. PMID 15951544
- [Derived] Stremmel W, Braun A, Hanemann A, Ehehalt R, Autschbach F, Karner M. Delayed release phosphatidylcholine in chronic-active ulcerative colitis: a randomized, double-blinded, dose finding study. J Clin Gastroenterol. 2010 May-Jun;44(5):e101-7. doi: 10.1097/MCG.0b013e3181c29860. PMID 20048683